CLINICAL TRIAL: NCT01809262
Title: Single Dose Preliminary Dose-ranging and Safety in Patients With COPD
Brief Title: Single Dose Ranging Study of BI 1744 CL (Olodaterol) in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.3
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (6):
- olodaterol 2 mcg (Experimental): solution for inhalation
  Interventions: Drug: single dose of 2 mcg
- olodaterol 5 mcg (Experimental): solution for inhalation
  Interventions: Drug: single dose of 5 mcg
- olodaterol 10 mcg (Experimental): solution for inhalation
  Interventions: Drug: single dose of 10 mcg
- olodaterol 20 mcg (Experimental): solution for inhalation
  Interventions: Drug: single dose of 20 mcg
- olodaterol 40 mcg (Experimental): solution for inhalation
  Interventions: Drug: single dose of 40 mcg
- placebo (Placebo Comparator): solution for inhalation
  Interventions: Drug: single dose of placebo

INTERVENTIONS:
Drug: single dose of 5 mcg — solution for inhalation
  Arms: olodaterol 5 mcg
Drug: single dose of placebo — solution for inhalation
  Arms: placebo
Drug: single dose of 40 mcg — solution for inhalation
  Arms: olodaterol 40 mcg
Drug: single dose of 20 mcg — solution for inhalation
  Arms: olodaterol 20 mcg
Drug: single dose of 2 mcg — solution for inhalation
  Arms: olodaterol 2 mcg
Drug: single dose of 10 mcg — solution for inhalation
  Arms: olodaterol 10 mcg

SUMMARY:
Primary objective: To investigate bronchodilator effect and safety of single doses of BI 1744 CL inhaled via Respimat inhaler, Secondary objective: to characterize pharmacokinetics of BI 1744 CL. Olodaterol dose 40 mcg was investigated only in the open-label extension part for additional PK assessments which are not defined as primary or secondary endpoints.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease
2. Smoking history of more than 10-pack years

Exclusion criteria:

1. History of asthma, allergic rhinitis, myocardial infarction or unstable of life-threatening cardiac arrhythmias
2. Marked baseline prolongation of QT/QTc interval

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1222.3.1 Atrium medisch centrum, Heerlen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Pharmacokinetic sub-study to characterise the pharmacokinetics of 2 μg to 20 μg Olodaterol was planned in a subset of 18 patients. After preliminary evaluation of the data, an open-label extension was planned to investigate the safety, tolerability, and pharmacokinetics of single doses of 40 μg Olodaterol in the 18 patients of the PK sub-study.
Pre-assignment Details: This was a randomised, Double-Blind, Placebo-Controlled, 5-Way crossover trial. Each treatment was only administered once in a single dose with a washout period of at least 14 days between treatments.
Groups:
- Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg: Patients were administered matching Placebo in the first period, Olodaterol 2 mcg qd in the second period, Olodaterol 20 mcg qd in the third period, Olodaterol 5 mcg qd in the fourth period and Olodaterol 10 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg: Patients were administered matching Placebo in the first period, Olodaterol 20 mcg qd in the second period, Olodaterol 2 mcg qd in the third period, Olodaterol 10 mcg qd in the fourth period and Olodaterol 5 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg: Patients were administered Olodaterol 2 mcg qd in the first period, Olodaterol 5 mcg qd in the second period, matching Placebo in the third period, Olodaterol 10 mcg qd in the fourth period and Olodaterol 20 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg: Patients were administered Olodaterol 2 mcg qd in the first period, matching Placebo in the second period, Olodaterol 5 mcg qd in the third period, Olodaterol 20 mcg qd in the fourth period and Olodaterol 10 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 2 mcg qd in the second period, Olodaterol 10 mcg qd in the third period, matching Placebo in the fourth period and Olodaterol 20 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 10 mcg qd in the second period, Olodaterol 2 mcg qd in the third period, Olodaterol 20 mcg qd in the fourth period and matching Placebo in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 20 mcg qd in the second period, Olodaterol 5 mcg qd in the third period, matching Placebo in the fourth period and Olodaterol 10 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 5 mcg qd in the second period, Olodaterol 20 mcg qd in the third period, Olodaterol 2 mcg qd in the fourth period and matching Placebo in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg: Patients were administered Olodaterol 20 mcg qd in the first period, matching Placebo in the second period, Olodaterol 10 mcg qd in the third period, Olodaterol 2 mcg qd in the fourth period and Olodaterol 5 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg: Patients were administered Olodaterol 20 mcg qd in the first period, Olodaterol 10 mcg qd in the second period, matching Placebo in the third period, Olodaterol 5 mcg qd in the fourth period and Olodaterol 2 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
Period: Period 1 (First Dose + Washout)
Arm/Group | Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg | Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg | Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg | Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo | Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg | Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo | Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg | Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg
Started | 4 | 4 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Second Dose + Washout)
Arm/Group | Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg | Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg | Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg | Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo | Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg | Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo | Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg | Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg
Started | 4 | 4 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Third Dose + Washout)
Arm/Group | Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg | Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg | Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg | Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo | Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg | Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo | Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg | Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg
Started | 4 | 4 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (Fourth Dose + Washout)
Arm/Group | Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg | Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg | Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg | Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo | Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg | Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo | Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg | Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg
Started | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5 (Fifth Dose + Washout)
Arm/Group | Placebo / Olo 2mcg / Olo 20mcg / Olo 5mcg / Olo 10mcg | Placebo / Olo 20mcg / Olo 2mcg / Olo 10mcg / Olo 5mcg | Olo 2mcg / Olo 5mcg / Placebo / Olo 10mcg / Olo 20mcg | Olo 2mcg / Placebo / Olo 5mcg / Olo 20mcg / Olo 10mcg | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 5mcg / Olo 10mcg / Olo 2mcg / Olo 20mcg / Placebo | Olo 10mcg / Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg | Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg / Placebo | Olo 20mcg / Placebo / Olo 10mcg / Olo 2mcg / Olo 5mcg | Olo 20mcg / Olo 10mcg / Placebo / Olo 5mcg / Olo 2mcg
Started | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 4 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: Total number of patients treated in the study. This was a double-blind, 5-period crossover trial. Each of the 36 patients received placebo and 4 single doses of Olodaterol (Olo) (2 microgram (mcg), 5 mcg, 10 mcg, 20mcg) separated by a wash-out period of at least 14 days.
Arm/Group | Study Total
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) at 24 Hours After a Single-dose of Study Treatment
Description: Forced expiratory volume in one second (FEV1) at 24 hours after a single-dose of study treatment. Means are adjusted with test-day baseline, patient, treatment, and period as fixed effects. Test-day baseline value was defined as the value at 10 minutes before inhalation of study medication.
Time Frame: 24 hours post-dosing
Population: Full Analysis Set (FAS): The FAS consisted of all treatment periods with baseline data and post-dosing data for FEV1 at 24 hours.
Measure: Mean (Standard Error); unit: L
Groups:
- Placebo: Single dose of matching placebo delivered by the Respimat inhaler.
- Olo 2 mcg: Single dose of Olodaterol 2 mcg delivered by the Respimat inhaler.
- Olo 5 mcg: Single dose of Olodaterol 5mcg delivered by the Respimat inhaler.
- Olo 10 mcg: Single dose of Olodaterol 10 mcg delivered by the Respimat inhaler.
- Olo 20 mcg: Single dose of Olodaterol 20 mcg delivered by the Respimat inhaler.
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 0.916 (0.014) | 0.986 (0.014) | 1.015 (0.014) | 1.029 (0.014) | 1.035 (0.014)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 0.070, 95% CI [0.031 to 0.109], Standard Error of Mean 0.020
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.099, 95% CI [0.060 to 0.138], Standard Error of Mean 0.020
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.113, 95% CI [0.074 to 0.152], Standard Error of Mean 0.020
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.119, 95% CI [0.080 to 0.158], Standard Error of Mean 0.020

2. Secondary Outcome: FEV1 AUC 0 - 3 Hours
Description: The FEV1 AUC was calculated as the area under the curve above zero as the horizontal axis from zero time to 3 hours, using the trapezoidal rule divided by 3 hours to give the results in litres. The test-day baseline (defined as the pulmonary function test (PFT) at 10 minutes before inhalation of study medication) was assigned to time zero.
Time Frame: -10 minutes (min), 30min, 1 hour (h), 2h and 3h post-dosing
Population: Full Analysis Set (FAS): The FAS consisted of all treatment periods with baseline data and post-dosing data available for this endpoint
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 0.997 (0.011) | 1.105 (0.011) | 1.152 (0.011) | 1.158 (0.011) | 1.189 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.108, 95% CI [0.077 to 0.139], Standard Error of Mean 0.016
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.155, 95% CI [0.124 to 0.186], Standard Error of Mean 0.016
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.161, 95% CI [0.130 to 0.192], Standard Error of Mean 0.016
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.192, 95% CI [0.161 to 0.223], Standard Error of Mean 0.016

3. Secondary Outcome: FEV1 AUC 0 - 12 Hours
Description: The FEV1 AUC was calculated as the area under the curve above zero as the horizontal axis from zero time to 12 hours, using the trapezoidal rule divided by 12 hours to give the results in litres. The test-day baseline (defined as the pulmonary function test (PFT) at 10 minutes before inhalation of study medication) was assigned to time zero.
Time Frame: -10 minutes (min), 30min, 1 hour (h), 2h, 3h, 4h, 6h, 8h, 10h and 12h post-dosing
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 0.954 (0.012) | 1.053 (0.011) | 1.093 (0.011) | 1.108 (0.012) | 1.138 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.099, 95% CI [0.068 to 0.131], Standard Error of Mean 0.016
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.139, 95% CI [0.107 to 0.171], Standard Error of Mean 0.016
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.153, 95% CI [0.122 to 0.185], Standard Error of Mean 0.016
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.184, 95% CI [0.152 to 0.215], Standard Error of Mean 0.016

4. Secondary Outcome: FEV1 AUC 0 - 24 Hours
Description: The FEV1 AUC was calculated as the area under the curve above zero as the horizontal axis from zero time to 24 hours, using the trapezoidal rule divided by 24 hours to give the results in litres. The test-day baseline (defined as the pulmonary function test (PFT) at 10 minutes before inhalation of study medication) was assigned to time zero.
Time Frame: -10 minutes (min), 30min, 1 hour (h), 2h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 22h, 23h and 24h post-dosing
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 0.923 (0.011) | 1.009 (0.011) | 1.040 (0.011) | 1.061 (0.011) | 1.085 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.087, 95% CI [0.056 to 0.117], Standard Error of Mean 0.015
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.118, 95% CI [0.087 to 0.148], Standard Error of Mean 0.015
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.138, 95% CI [0.107 to 0.168], Standard Error of Mean 0.015
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.162, 95% CI [0.132 to 0.193], Standard Error of Mean 0.015

5. Secondary Outcome: FEV1 AUC 12 - 24 Hours
Description: The FEV1 AUC was calculated as the area under the curve above zero as the horizontal axis from 12 hours to 24 hours, using the trapezoidal rule divided by 12 hours to give the results in litres. The test-day baseline (defined as the pulmonary function test (PFT) at 10 minutes before inhalation of study medication) was assigned to time zero.
Time Frame: 12h, 14h, 22h, 23h and 24h post-dosing
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 0.891 (0.012) | 0.965 (0.012) | 0.987 (0.012) | 1.014 (0.012) | 1.032 (0.012)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.074, 95% CI [0.041 to 0.108], Standard Error of Mean 0.017
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.096, 95% CI [0.062 to 0.130], Standard Error of Mean 0.017
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.122, 95% CI [0.089 to 0.156], Standard Error of Mean 0.017
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.141, 95% CI [0.107 to 0.174], Standard Error of Mean 0.017

6. Secondary Outcome: Peak FEV1 From 0 to 3 Hours
Description: Peak FEV1 was defined as the maximum values of FEV1 from 0 to 3 hours.
Time Frame: 0 to 3 hours post-dosing
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 1.043 (0.013) | 1.164 (0.013) | 1.209 (0.013) | 1.219 (0.014) | 1.256 (0.013)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.121, 95% CI [0.084 to 0.158], Standard Error of Mean 0.019
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.166, 95% CI [0.129 to 0.203], Standard Error of Mean 0.019
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.176, 95% CI [0.139 to 0.214], Standard Error of Mean 0.019
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.213, 95% CI [0.176 to 0.250], Standard Error of Mean 0.019

7. Secondary Outcome: Peak Forced Vital Capacity (FVC) From 0 to 3 Hours
Description: Peak FVC was defined as the maximum values of FVC from 0 to 3 hours.
Time Frame: 0 to 3 hours post-dosing
Population: as for outcome 2
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
L | 3.134 (0.035) | 3.440 (0.035) | 3.489 (0.035) | 3.485 (0.035) | 3.589 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 2 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.306, 95% CI [0.210 to 0.402], Standard Error of Mean 0.049
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.355, 95% CI [0.258 to 0.452], Standard Error of Mean 0.049
Statistical Analysis 3: Comparison: Placebo vs Olo 10 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.350, 95% CI [0.253 to 0.447], Standard Error of Mean 0.049
Statistical Analysis 4: Comparison: Placebo vs Olo 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.455, 95% CI [0.359 to 0.551], Standard Error of Mean 0.049

8. Secondary Outcome: Time to Peak Bronchodilator Response
Description: A bronchodilator response was considered to have been achieved if an FEV1 measurement of at least 12% greater than the test-day baseline value was recorded at any time during the first 3 hours of observation after dosing.
Time Frame: 0 to 3 hours post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
minutes | 102.0 (57.4) | 92.6 (55.1) | 98.6 (53.8) | 83.8 (46.6) | 96.9 (39.9)

9. Secondary Outcome: Time to Onset of Response
Description: Onset of the bronchodilator response after a single dose of study treatment was defined as the linear interpolation of the time of the first bronchodilator response and the time of the observation just prior to the first bronchodilator response (even if that is the baseline observation). If none of the FEV1 values in the first 3 hours after dosing exceeded 12% of the pre-dose value, then the onset was set to 3 hours plus 1 minute.
Time Frame: 0 to 3 hours post-dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
minutes | 148.9 (56.2) | 91.5 (73.6) | 57.5 (68.5) | 59.9 (69.6) | 38.2 (48.1)

10. Secondary Outcome: Number of Patients Requiring Rescue Medication on a Test-day
Description: Number of Patients Requiring Rescue Medication on a Test-day. Salbutamol inhalation aerosol MDI (Ventolin®, 100 μg/actuation) was provided for use as rescue medication. Administration of rescue medication can occur at any point during the pulmonary function testing as deemed necessary by the patient or the investigator.
Time Frame: Visits 1,2,4,5,6
Population: Safety set which consisted of all randomised patients who had taken at least one dose of study medication.
Measure: Number; unit: Number of Patients
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
Number of Patients | 4 | 4 | 0 | 1 | 1

11. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events (cardiac disorders and investigations).
Time Frame: 2 weeks
Population: Safety set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 35 | 35 | 35 | 34 | 35
percentage of participants
  Cardiac disorders | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased | 0.0 | 0.0 | 0.0 | 2.9 | 0.0

12. Secondary Outcome: Laboratory Testing: Average Change From Baseline of Potassium and Calcium
Description: Laboratory testing: Average change from baseline of potassium and calcium measured on test-days
Time Frame: Baseline and Visit 6
Population: Safety set.
Measure: Geometric Mean (Inter-Quartile Range); unit: mmol/L
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 18 | 18 | 17 | 17 | 18
mmol/L
  Potassium (N=17, 18, 17, 17, 18) | 1.03 (NA) [0.99 to 1.07] | 1.01 (NA) [0.98 to 1.03] | 0.99 (NA) [0.95 to 1.03] | 0.98 (NA) [0.97 to 1.02] | 0.97 (NA) [0.92 to 1.01]
  Calcium (N=18, 18, 17, 17, 18) | 1.02 (NA) [0.99 to 1.03] | 1.00 (NA) [0.99 to 1.03] | 1.00 (NA) [0.98 to 1.01] | 1.01 (NA) [1.00 to 1.03] | 1.01 (NA) [0.99 to 1.04]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Single dose including washout phase
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/35 | 2/35 | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 5/35 | 2/35 | 4/35 | 5/34 | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Olo 2 mcg (N=35) | Olo 5 mcg (N=35) | Olo 10 mcg (N=34) | Olo 20 mcg (N=35)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Olo 2 mcg (N=35) | Olo 5 mcg (N=35) | Olo 10 mcg (N=34) | Olo 20 mcg (N=35)
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No